CLINICAL TRIAL: NCT03391050
Title: A Phase Ib/II Study to Investigate the Safety and Clinical Activity of APR-246 in Combination With Dabrafenib in Patients With BRAF V600 Mutant Unresectable and/or mEtastatic Cutaneous MElanoma Resistant to Dabrafenib/Trametinib Combination
Brief Title: A Study of APR-246 in Combination With Dabrafenib in Resistant Patients With BRAF V600 Mutant Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Target patient population - difficult to find patientes
Sponsor: Aprea Therapeutics (Industry)
Collaborators: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APR-633
Record Dates: First submitted 2017-12-19; First posted 2018-01-05 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Melanoma
Keywords: Melanoma; Malignant melanoma; Skin cancer; Resistant cancer; Unresectable cancer; Metastatic cancer; BRAF mutant
MeSH Terms: conditions — Melanoma; Skin Neoplasms; Neoplasm Metastasis | interventions — eprenetapopt; dabrafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- APR-246 + Dabrafenib (Experimental)
  Interventions: Drug: APR-246; Drug: Dabrafenib

INTERVENTIONS:
Drug: APR-246 — Intravenous infusion
Drug: Dabrafenib — Oral administration

SUMMARY:
The purpose of this study is to make a preliminary assessment of the efficacy of a combined APR-246 and dabrafenib therapy regimen in patients with BRAFV600 mutant unresectable and/or metastatic cutaneous melanoma resistant to the dabrafenib/trametinib combination. In addition, the study aims to assess the safety profile of the combined APR-246 and dabrafenib therapy regimen, to explore potential biomarkers, and to further describe the anti-tumour activity of the combination of APR-246 and dabrafenib. The trial will enroll up to 31 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed BRAF V600 mutation-positive unresectable and/or metastatic malignant cutaneous melanoma, as determined locally by a validated test and treated with dabrafenib/trametinib first line combination therapy or second line after first line immunotherapy.
* Patients that have progressed according to RECIST 1.1 after at least 4 weeks of treatment with dabrafenib/trametinib and remained on dabrafenib full dose (150mg bid) treatment for the study.
* Measurable disease according to RECIST 1.1 criteria. For phase II only, metabolic measurable disease (according to PERCIST).
* Availability of tissue from a metastatic lesion. A new biopsy is required unless inaccessible. An archival sample is accepted in that case after discussion with the sponsor.
* ECOG Performance Status of 0 or 1.
* Patients able to swallow and retain oral medication.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* For female patients of childbearing potential, a pregnancy test (serum) will be performed within 7 days before inclusion. Woman of childbearing potential must be willing to use one highly effective form of contraception during anticancer treatment and for at least six months thereafter. Men must agree to use condom during the course of this study and at least six months after the last administration of the study treatment and contraception should be considered for partner of childbearing potential.
* Adequate organ system function.
* Signed informed consent before any study specific procedure and/or treatment happens.

Exclusion Criteria:

* Presence of uveal melanoma and/or other non-cutaneous melanomas.
* Current use of a prohibited medication or need for any of these medications during treatment with study drug and within 28 days before the first administration of APR-246. I.e., no anti-cancer other than that given in this clinical trial, no immunotherapy, no hormonal cancer therapy, no radiation therapy (except palliative) and no experimental medications are permitted during the trial. All alternative therapies must first be approved by the sponsor. Supportive care therapies are allowed.
* Unresolved toxicity greater than NCI-CTCAE(v4) Grade 1 from previous anti-cancer therapy except alopecia.
* Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of drugs.
* Known HIV, active hepatitis B or hepatitis C infection.
* Primary malignancy of the central nervous system.
* History of familial long QT, serious ventricular arrhythmia (no VT > 130 bpm and > 5 extra beats per minute), no QTc ≥ 480 msec calculated from a single ECG reading or a mean of 3 ECG readings using Fridericia's correction (QTcF = QT/RR0.33) or bradycardia (< 45 bpm).
* Untreated or symptomatic brain metastasis, leptomeningeal disease or spinal cord compression. Patients who are on a stable dose of corticosteroids > 1 month or off corticosteroids for 2 weeks can be enrolled.
* History of acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting, or thrombo-embolic event within the past 24 weeks from signature of ICF.
* Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drugs, or excipients.
* Uncontrolled diabetes, hypertension or other medical conditions that may interfere with assessment of toxicity.
* Pregnant or lactating woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
Phase Ib: Adverse Events (AEs) | Up to 30 days after last study treatment day, or at end of study visit due to progression, whichever occurs later (treatment cycles are stopped due to progression, toxicity or patient's decision)
  Clinical and laboratory adverse events (AEs) and serious adverse events (SAEs) will be reported and graded
Phase Ib: Dose Limiting Toxicities (DLTs) | Until end of cycle 1 (cycle length is 28 days)
Phase II: Objective response rate by RECIST1.1 | Until progression (assessed up to 12 months)

SECONDARY OUTCOMES:
Clinical benefit rate | Until progression (assessed up to 12 months)
  Proportion of patients with a CR, PR or Stable Disease (SD) ≥ 4 months
Duration of response | Until progression (assessed up to 12 months)
Progression free survival (PFS) | Until progression (assessed up to 12 months)
Area under the plasma concentration versus time curve (AUC) for APR-246 | Until Cycle 1 Day 8 (Phase Ib) or Cycle 1 Day 1 (Phase II)
Plasma drug concentration at a specified time t (Ct) for APR-246 | Until Cycle 1 Day 8 (Phase Ib) or Cycle 1 Day 1 (Phase II)
Maximum observed plasma concentration (Cmax) of APR-246 | Until Cycle 1 Day 8 (Phase Ib) or Cycle 1 Day 1 (Phase II)
Time to reach maximum plasma concentration following drug administration (tmax) for APR-246 | Until Cycle 1 Day 8 (Phase Ib) or Cycle 1 Day 1 (Phase II)
Assessment of metabolic response | Until Cycle 2 Day 1 (cycle length is 28 days)
  According to classical PERCIST criteria (30%) modified PERCIST criteria (15%) and the consistency classification

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Awada, PhD, Study Chair — Jules Bordet Institute, Brussels, Belgium; Joseph Kerger, MD, Principal Investigator — Jules Bordet Institute, Brussels, Belgium
Locations (3):
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - CHU UCL Namur - site Sainte-Elisabeth, Namur

REFERENCES:
- [Background] Lehmann S, Bykov VJ, Ali D, Andren O, Cherif H, Tidefelt U, Uggla B, Yachnin J, Juliusson G, Moshfegh A, Paul C, Wiman KG, Andersson PO. Targeting p53 in vivo: a first-in-human study with p53-targeting compound APR-246 in refractory hematologic malignancies and prostate cancer. J Clin Oncol. 2012 Oct 10;30(29):3633-9. doi: 10.1200/JCO.2011.40.7783. Epub 2012 Sep 10. PMID 22965953
- [Background] Deneberg S, Cherif H, Lazarevic V, Andersson PO, von Euler M, Juliusson G, Lehmann S. An open-label phase I dose-finding study of APR-246 in hematological malignancies. Blood Cancer J. 2016 Jul 15;6(7):e447. doi: 10.1038/bcj.2016.60. No abstract available. PMID 27421096
- See also: Aprea Therapeutics AB's website (Sponsor) — http://www.aprea.com/